CLINICAL TRIAL: NCT03910764
Title: Retrospective Surveillance Study of Candiduria in Hospitalized Patients
Brief Title: Surveillance Study of Candiduria in Hospitalized Patients
Status: Completed | Type: Observational
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Chen Ying-Chun, infection preventionist, Taichung Veterans General Hospital
Other Study IDs: CE18273B
Record Dates: First submitted 2019-04-07; First posted 2019-04-10 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-10

CONDITIONS: Candiduria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: no intervention — Investigators review patients' medical records and collect personal data, underlying diseases, indwelling catheter duration, laboratory data, diagnosis, treatment and prognosis.

SUMMARY:
The purpose of the study is to explore the epidemiology, underlying diseases, indwelling catheter duration, laboratory data, diagnosis, treatment and prognosis of patients with Candiduria.

DETAILED DESCRIPTION:
The study is a retrospective study. Investigators will review medical records of patients with Candiduria from January 2015 to December 2017 to collect data about personal data, underlying diseases, indwelling catheter duration, laboratory data of urine routines and urine cultures, the symptom of fever, diagnosis, treatment and prognosis. After the data collection, investigators will run a descriptive statistics to find out the profile of the medical care of Candiduria in Taiwan.

ELIGIBILITY:
Inclusion Criteria:

* patients with Candiduria

Exclusion Criteria:

* patients without Candiduria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: all patients with Candiduria
Sampling Method: Non-Probability Sample
Enrollment: 536 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
prevalence rate of Candiduria | January 2015 to December 2017
  the number of patients with Candiduria/ the number of all hospitalized patients
morbidity rate of underlying diseases | January 2015 to December 2017
  the proportion of patients with every specific underlying disease
indwelling catheter rate | January 2015 to December 2017
  the proportion of patients with indwelling catheter
pyuria rate | January 2015 to December 2017
  the proportion of patients with pyuria
Candiduria rate | January 2015 to December 2017
  the proportion of patients with Candiduria
treatment rate | January 2015 to December 2017
  the proportion of patients with Candiduria treated with antifungal agents
mortality rate | January 2015 to December 2017
  1. the number of patients who die / the number of all hospitalized patients
  2. the number of patients who die from Candiduria/ the number of all hospitalized patients
average indwelling catheter duration | January 2015 to December 2017
  The sum of indwelling catheter durations / the number of all hospitalized patients with Candiduria

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No